CLINICAL TRIAL: NCT01174602
Title: Randomized Controlled Trial of Inpatient Exposure Therapy and Response Prevention for Anorexia Nervosa
Brief Title: Inpatient Exposure Therapy and Response Prevention & Cognitive Remediation Therapy for Anorexia Nervosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); National Alliance for Research on Schizophrenia and Depression (Other); The Hilda & Preston Davis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6010; 1R01MH082736-01 (NIH)
Record Dates: First submitted 2010-07-29; First posted 2010-08-03 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa | interventions — Implosive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exposure Therapy for AN (AN-EX/RP) (Experimental): Exposure Therapy and Ritual Prevention (AN-EX/RP) includes 12 sessions of confronting feared eating situations without the use of anxiety reducing behaviors.
  Interventions: Behavioral: Exposure Therapy for AN (AN-EX/RP)
- Cognitive Remediation Therapy (Active Comparator): Cognitive Remediation Therapy (CRT)
  Interventions: Behavioral: Cognitive Remediation Therapy

INTERVENTIONS:
Behavioral: Exposure Therapy for AN (AN-EX/RP) — 12 Sessions, 3 times per week. 90 minute sessions. Group therapy twice per week.
  Arms: Exposure Therapy for AN (AN-EX/RP)
Behavioral: Cognitive Remediation Therapy — 12 Sessions, 3 times per week. 45 minute sessions. Group therapy twice per week.
  Arms: Cognitive Remediation Therapy

SUMMARY:
Exposure and response prevention (AN-EXRP) will help individuals with anorexia nervosa improve their eating behavior.

DETAILED DESCRIPTION:
Anorexia nervosa (AN) is a serious illness associated with substantial morbidity and a mortality rate among the highest of any psychiatric illness. The rate of relapse is disturbingly high, with up to 50% of patients requiring re-hospitalization within a year of discharge. Current treatments are inadequate in helping older adolescents and adults achieve sustained recovery. Importantly, eating behavior remains disturbed after weight restoration: patients demonstrate restrictive eating in their self-selected foods and in standardized meals, and caloric intake in standardized meals is inversely related to pre-meal anxiety. Emerging data suggest that eating behavior is particularly important in post-hospital course, and that significantly altering eating behavior is critical in improving outcome for these individuals. Furthermore, caloric intake in standardized meals has been shown to be related to pre-meal anxiety. This study evaluates the potential utility of two psychotherapeutic interventions in improving eating behavior prior to hospital discharge. Each individual receives, in random order, Cognitive Remediation Therapy for 4 weeks and Exposure and Response Prevention for AN for 4 weeks. The investigators hypothesize that these interventions will lead to improvement in eating behavior, measured by food diaries and standardized meals.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-IV-TR™ diagnosis of anorexia nervosa (restricting or binge-purge subtype), with or without amenorrhea at the time of inpatient admission
2. Subjects will have achieved 85% of ideal body weight (IBW)
3. Age 16-45 years
4. No acute medical condition
5. Subjects must have signed informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

1. Psychotic or bipolar I disorder
2. Substance abuse or dependence in the last 6 months
3. Current Axis I disorder requiring psychotropic medication (ongoing antidepressant treatment for stable comorbid conditions will be allowed)
4. Significant co-morbid depression
5. Significant medical problems that would introduce additional risk related to research or interfere with participation, e.g. SBP>140, DBP>90, HR>100 for a sustained period.
6. Active suicidal intent

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2009-11; Primary Completion 2011-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Eating Behavior | 4 weeks
  Eating behavior will be measured as both intake patterns in food records and in a laboratory based meal.

SECONDARY OUTCOMES:
Psychological Improvement | 4 weeks
  The impact of these interventions on psychological state, including anxiety and thinking patterns, will be measured.
Psychological Improvement | 8 weeks
  The impact of these interventions on psychological state, including anxiety and thinking patterns, will be measured.
Eating Behavior | 8 weeks
  Laboratory meal after crossover condition.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Steinglass, MD, Principal Investigator — NYSPI
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States